CLINICAL TRIAL: NCT04484285
Title: Home Operations Utilizing Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201901518 -A
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Performance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Younger Cohort (Active Comparator): Healthy individuals aged 18 - 55
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation (tVNS)
- Older Cohort (Active Comparator): Healthy individuals aged 56 - 85
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation (tVNS)

INTERVENTIONS:
Device: Transcutaneous Vagal Nerve Stimulation (tVNS) — vagal nerve stimulation

SUMMARY:
This project will utilize a home-operated stimulator in 1) a healthy young adult population and 2) a healthy older adult population to provide a proof of concept of home-use of transcutaneous vagal nerve stimulation (tVNS). tVNS is believed to modulate cognitive performance.

DETAILED DESCRIPTION:
The vagal nerve is a major component of the autonomic nervous system and mediates the physiological responses of major organs during moments of stress and learning, including brain areas that modulate cognitive performance. Vagal nerve stimulation (VNS) has been indicated to improve stress response and to enhance neuroplasticity by directly impacting brain structures critical for cognition. Historically, VNS methods required neurosurgery and were reserved for medically intractable epilepsy or other severe conditions. Today, vagal nerve stimulation can be performed with a minimal-risk non-invasive approach without surgery through a technique called transcutaneous Vagal Nerve Stimulation (tVNS). This project will utilize a home-operated stimulator in healthy young adult and healthy older populations to provide a proof of concept of practical home-use stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Participants for one cohort will be adults between the ages of 18-55, consistent with the typical college population
* Participants for the other cohort will be adults between the ages of 56 - 85. Participants must read and write English.

Exclusion Criteria:

* Major medical illnesses including diagnosed severe neurological illnesses (e.g., stroke, seizure history), autoimmune disorders, and severe psychiatric diseases (e.g., schizophrenia) will be excluded. Participants with any history of brain surgery, tumor, intracranial metal implantation, pacemakers or other implanted devices will be excluded.
* Sleep medications and/or psychostimulants are exclusionary. Subjects in the older cohort will NOT be excluded for taking blood pressure and cholesterol medication. Participants who are pregnant will be excluded. If participants have a history of adverse reaction to electrical nerve stimulation, they will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida McKnight Brain Institute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Younger Cohort: Healthy individuals aged 18 - 50
  Transcutaneous Vagal Nerve Stimulation (tVNS): vagal nerve stimulation completed at home for 7 days.
- Older Cohort: Healthy individuals aged 50 - 85
  Transcutaneous Vagal Nerve Stimulation (tVNS): vagal nerve stimulation completed at home for 7 days.
Period: Overall Study
Arm/Group | Younger Cohort | Older Cohort
Started | 9 | 1
Completed | 6 | 1
Not Completed | 3 | 0
Not completed — Unable to operate stimulator | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Younger Cohort: Healthy individuals aged 18 - 50
  Transcutaneous Vagal Nerve Stimulation (tVNS): vagal nerve stimulation
- Older Cohort: Healthy individuals aged 50 - 85
  Transcutaneous Vagal Nerve Stimulation (tVNS): vagal nerve stimulation
- Total: Total of all reporting groups
Arm/Group | Younger Cohort | Older Cohort | Total
Number analyzed (Participants) | 9 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 1 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 9 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 1 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale
Description: This is a standard version of a usability scale. Subjects will be given 10 statements regarding the usability of the equipment they used, and they will report how much they agree with each statement on a 1 - 5 scale (1 is strongly disagree and 5 is strongly agree). The score range is 10-50 where 50 demonstrates the highest acceptance of the usability of the device and 10 demonstrates the lowest acceptance of the usability of the device.
Time Frame: Day 7 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Younger Cohort | Older Cohort
Number analyzed (Participants) | 6 | 1
score on a scale | 46.25 (18.53) | 10 (NA) — Standard Deviation not calculated for one participant

ADVERSE EVENTS:
Time Frame: 7 days
Description: The study intervention utilized a stimulator designed for home use. This design has additional hardware and software features that reduces the chance of and adverse event. On the hardware, the device runs off 4 double AA batteries opposed to plugged into an outlet. On software, initiation of the device is dependent on the corresponding web portal which is programmed to limit use duration per session and to one session per day.
Arm/Group | Younger Cohort | Older Cohort
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/1
Other Adverse Events (participants affected / at risk) | 0/9 | 0/1

LIMITATIONS AND CAVEATS:
The study enrolled only participant into the older adult group. This participant was unable to use the stimulator. To understand the feasibility of this intervention in this group many more older adult participants would need to be enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04484285/Prot_SAP_002.pdf
  • Informed Consent Form (2020-07-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04484285/ICF_003.pdf